CLINICAL TRIAL: NCT02330237
Title: Safety and Efficacy of Natural Gel Combination and Hair Mask of Plant Origin in Patients With Psoriasis: A Randomized, Double-Blind, Placebo (Vehicle) Controlled
Brief Title: Natural Gels for Treatment of Plaque Psoriasis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Secret of Youth (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NGCPP
Record Dates: First submitted 2014-12-30; First posted 2015-01-01 (Estimated); Last update posted 2018-07-23 (Actual); Status verified 2018-07

CONDITIONS: Parapsoriasis
MeSH Terms: conditions — Parapsoriasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- patients (Active Comparator): natural gels
  Interventions: Drug: natural gels
- subjects (Placebo Comparator): These patients will receive that placebo (vehicle) products.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: natural gels — whole fruits and vegetables
  Other Names: plant origin
  Arms: patients
Drug: Placebo
  Arms: subjects

SUMMARY:
The aim of the study is to evaluate the safety and the therapeutic activity of the combination of Natural Gel combination and hair mask of plant origin in patients with mild to moderate plaque psoriasis.

DETAILED DESCRIPTION:
This is a random, double blind placebo -vehicle- controlled study. Patients recruiting and inclusion into the study is well defined. Expert on site monitoring will assure execution of all assignments as detailed in the protocol (screening, consent form, double-blind group assignment) .

Statistical analysis:

* It is calculated that 52 patients will be needed for this study.
* Type I error probability associated with this test is 0.05 .
* Uncorrected chi square will be used to assess changes in the measured variables.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with stable (for at least 6 months), mild to moderate (less than 10% of the skin surface area) plaque psoriasis.
2. Male and female ≥ 18 years old.
3. Subject is capable of giving a written informed consent.

Exclusion Criteria:

1. Subjects treated by topical or photo or systemic anti psoriatic therapy during 4 weeks prior to the study.
2. Subjects treated with Biological products for psoriasis for the last 3 months prior to starting the present study.
3. Subjects with any other type of psoriasis but vulgaris (plaque ).
4. Use of investigational agents < 30 days prior to the study.
5. Low compliance.
6. Subjects who are mentally or physically unable to comply with all aspects of the study.
7. Pregnant women.
8. Known allergic reaction to fragrance or any ingredient of the test products.
9. Other inflammatory skin disease in the treatment area that may confound the evaluation of the psoriasis.
10. A medical condition that may put the patient at a general risk and therefore would prevent participation in the clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2015-01; Primary Completion 2016-11 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Modified Psoriasis Assessment severity index | up to 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Felix Pavlotzky, MD, Principal Investigator — Chaim sheba Medical Center, Dept. of Dermatolgy. Tel-Hashomer, Israel
Locations (1):
- Chaim Sheba Med. center. Dept. Of Dermatology, Reamat- Gan, Ramat-almogi, Israel